CLINICAL TRIAL: NCT04032301
Title: Characterization of Comorbid Post-traumatic Stress Disorder and Major Depressive Disorder Utilizing Ketamine as an Experimental Medicine Probe
Brief Title: Repeated Ketamine Infusions for Comorbid PTSD and MDD in Veterans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PSYCH-2019-28086
Record Dates: First submitted 2019-06-26; First posted 2019-07-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Post-Traumatic Stress Disorders; Major Depressive Disorder
Keywords: ketamine; stress disorders, post-traumatic; stress disorders, traumatic; anxiety disorders; mental disorders; adjuvants, anesthesia; analgesics; anesthetics; anesthetics, dissociative; anesthetics, general; anesthetics, intravenous; excitatory amino acid agents; excitatory amino acid antagonists; hypnotics and sedatives; molecular mechanisms of pharmacological action; neurotransmitter agents; peripheral nervous system agents; pharmacologic actions; physiological effects of drugs; psychotropic drugs; sensory system agents; central nervous system agents; central nervous system depressants; depression; depressive disorder; depressive disorder, treatment-resistant; behavioral symptoms; mood disorders; therapeutic uses
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Stress Disorders, Traumatic; Anxiety Disorders; Mental Disorders; Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant; Behavioral Symptoms; Mood Disorders | interventions — Ketamine; Saline Solution; Sodium Chloride; Water

STUDY DESIGN:
Intervention Model Description: Experimental versus Placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous ketamine infusions (Experimental): Six infusions of 0.5 mg/kg ketamine hydrochloride solution over 3 weeks.
  Interventions: Drug: Ketamine
- Intravenous saline infusions (Placebo Comparator): Six infusions of normal saline solution over 3 weeks.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Ketamine — Six infusions of intravenous 0.5 mg/kg ketamine hydrochloride solution over 3 weeks.
  Other Names: Ketamine Hydrochloride
  Arms: Intravenous ketamine infusions
Other: Normal Saline — Six infusions of intravenous normal saline solution over 3 weeks.
  Other Names: Sodium Chloride in Water
  Arms: Intravenous saline infusions

SUMMARY:
Co-occurring post-traumatic stress disorder (PTSD) and major depressive disorder (MDD) is the most common response to trauma; it is associated with poor clinical outcomes and substantial human disability. Veterans with both PTSD and MDD (PTSD+MDD) have been shown to be at much greater suicidal risk than individuals with only one of these disorders. Ketamine given as repeated infusions has been shown to be effective in rapidly reducing PTSD and MDD symptoms in treatment resistant PTSD+MDD individuals. However, knowledge about the mechanisms underlying comorbid PTSD and MDD remain limited. The purpose of this study is to use repeated ketamine infusions as a probe to validate a model of PTSD+MDD that focuses on neuroanatomy and executive functioning.

DETAILED DESCRIPTION:
This study is designed to better characterize the neurocognitive and associated functional connectivity mechanisms underlying comorbid post-traumatic stress disorder (PTSD) and major depressive disorder (MDD) among veterans. Participants will be male/female veterans (18 to 75 years old) of any era or military background who suffer from chronic PTSD and MDD. Potential participants will be recruited from mental health clinics and screened for eligibility using a two stage process (phone/chart review, followed by interview). Participants with PTSD+MDD will undergo a series of baseline assessments including a baseline functional magnetic resonance imaging (fMRI) then be randomized to receive either 6 ketamine or 6 normal saline infusions on a Monday-Friday schedule over 3 weeks. On the day of infusion, participants will be required to stay at the clinical site for 2 hours after the infusion has been given. They will also be monitored via a phone call on the following day. After the infusion period has been completed participants will undergo a follow-up fMRI then 4 follow-up visits, up to 2 months. Additional participants will be enrolled in healthy control, depression only, and PTSD only groups and will only undergo baseline assessments, including a single fMRI.

ELIGIBILITY:
Inclusion Criteria:

For the PTSD+MDD group, inclusion criteria are:

1. Female/Male veterans
2. 18 to 75 years old
3. Meets DSM-5 criteria for MDD, single or recurrent, moderate-severe without psychotic features
4. Meets DSM-5 criteria for chronic PTSD or subthreshold PTSD [meets criterion A (traumatic event), criterion B (intrusion symptoms), and 2 of the following 3 criteria: C (avoidance symptoms), D (negative alterations in cognitions and mood), or E (marked alterations in arousal and reactivity)]
5. If applicable, 6 weeks of stable antidepressants/augmenting agents
6. Sixth grade reading level
7. Ability to provide consent

For the Healthy Controls group, inclusion criteria are:

1. Female/Male veterans
2. 18 to 75 years old
3. Does not meet DSM-5 criteria for MDD, single or recurrent, moderate-severe without psychotic features
4. Does not meet DSM-5 criteria for chronic PTSD or subthreshold PTSD
5. Not on medications for managing a psychiatric indication
6. Sixth grade reading level
7. Ability to provide consent

For the Depression-only group, inclusion criteria are:

1. Female/Male veterans
2. 18 to 75 years old
3. Experienced a traumatic event that meets DSM-5 criterion A for a diagnosis of PTSD but does not meet sufficient criteria (B-E) necessary for a diagnosis of PTSD or subthreshold PTSD
4. Meets criteria for MDD, single or recurrent, moderate-severe
5. If applicable, 6 weeks of stable antidepressants/augmenting agents
6. Sixth grade reading level
7. Ability to provide consent

For the PTSD-only group, inclusion criteria are:

1. Female/Male veterans
2. 18 to 75 years old
3. Meets DSM-5 criteria for chronic PTSD or subthreshold PTSD [meets criterion A (traumatic event), criterion B (intrusion symptoms), and 2 of the following 3 criteria: C (avoidance symptoms), D (negative alterations in cognitions and mood), or E (marked alterations in arousal and reactivity)]
4. Does not meet DSM-5 criteria for MDD, single or recurrent, moderate-severe without psychotic features
5. If applicable, 6 weeks of stable antidepressants/augmenting agents
6. Sixth grade reading level
7. Ability to provide consent

Exclusion Criteria:

For the PTSD+MDD group, exclusion criteria are:

1. Inability or unwillingness to provide written informed consent
2. Moderate/severe cognitive impairment
3. Current or lifetime diagnosis of psychosis-related disorder, bipolar I or II disorder, substance-induced mood disorder, or any mood disorder due to a general medical condition
4. History of moderate or severe traumatic brain injury
5. History of comorbid substance disorder within 1 month of screening
6. Prior use of ketamine as an antidepressant
7. Clinically unstable medical illness
8. For women: pregnancy (confirmed by baseline lab test), the initiation of female hormonal treatments within 3 months of screening, or inability or unwillingness to use a medically accepted contraceptive method for the duration of the study
9. Imminent risk of suicidal/homicidal ideation and/or behavior
10. Inability to undergo MRI (i.e. claustrophobia, ferromagnetic implants, etc.)

For the Healthy Controls group, exclusion criteria are:

1. Inability or unwillingness to provide written informed consent
2. Moderate/severe cognitive impairment
3. History of any major medical or psychiatric disorders
4. Current or lifetime diagnosis of psychosis-related disorder, bipolar I or II disorder, substance-induced mood disorder, or any mood disorder due to a general medical condition
5. History of moderate or severe traumatic brain injury
6. History of comorbid substance disorder within 1 month of screening
7. Prior use of ketamine as an antidepressant
8. Clinically unstable medical illness
9. For women: pregnancy (confirmed by baseline lab test), the initiation of female hormonal treatments within 3 months of screening, or inability or unwillingness to use a medically accepted contraceptive method for the duration of the study
10. Imminent risk of suicidal/homicidal ideation and/or behavior
11. Inability to undergo MRI (i.e. claustrophobia, ferromagnetic implants, etc.)

For the Depression-only group, exclusion criteria are:

1. Inability or unwillingness to provide written informed consent
2. Moderate/severe cognitive impairment
3. Meet DSM-5 criteria for PTSD or subthreshold PTSD
4. Current or lifetime diagnosis of psychosis-related disorder, bipolar I or II disorder, substance-induced mood disorder, or any mood disorder due to a general medical condition
5. History of moderate or severe traumatic brain injury
6. History of comorbid substance disorder within 1 month of screening
7. Prior use of ketamine as an antidepressant
8. Clinically unstable medical illness
9. For women: pregnancy (confirmed by baseline lab test), the initiation of female hormonal treatments within 3 months of screening, or inability or unwillingness to use a medically accepted contraceptive method for the duration of the study
10. Imminent risk of suicidal/homicidal ideation and/or behavior
11. Inability to undergo MRI (i.e. claustrophobia, ferromagnetic implants, etc.)

For the PTSD-only group, exclusion criteria are:

1. Inability or unwillingness to provide written informed consent
2. Moderate/severe cognitive impairment
3. Meet DSM-5 criteria for a diagnosis of MDD, single or recurrent, moderate to severe
4. Current or lifetime diagnosis of psychosis-related disorder, bipolar I or II disorder, substance-induced mood disorder, or any mood disorder due to a general medical condition
5. History of moderate or severe traumatic brain injury
6. History of comorbid substance disorder within 1 month of screening
7. Prior use of ketamine as an antidepressant
8. Clinically unstable medical illness
9. For women: pregnancy (confirmed by baseline lab test), the initiation of female hormonal treatments within 3 months of screening, or inability or unwillingness to use a medically accepted contraceptive method for the duration of the study
10. Imminent risk of suicidal/homicidal ideation and/or behavior
11. Inability to undergo MRI (i.e. claustrophobia, ferromagnetic implants, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | At baseline, 60 minutes pre-infusion, 24 hours post-infusion, and after infusion series up to 2 months.
  Change in major depressive disorder symptoms over the course of the intervention.
PTSD Symptom Scale-Interview for DSM-5 (PSS-I-5) | At baseline, 60 minutes pre-infusion, 24 hours post-infusion, and after infusion series up to 2 months.
  Change in post-traumatic stress disorder symptoms over the course of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina S Albott, MD, MA, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis Veterans Affairs Health Care System, Minneapolis, Minnesota, United States